CLINICAL TRIAL: NCT05889741
Title: Combining Stellate Ganglion Block With Prolonged Exposure for PTSD: A Randomized Clinical Trial
Brief Title: Combining Stellate Ganglion Block With Prolonged Exposure for PTSD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC20230087H
Record Dates: First submitted 2023-04-17; First posted 2023-06-05 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: SGB; Military
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The clinical staff, research staff, and the participant will be blind to study condition until after the 1-month follow-up assessment. After which time, the blind will be broken, and participants in the control condition will be offered the SGB.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Stellate Ganglion Block (Experimental): One time administration of a stellate ganglion block
  Interventions: Drug: Ropivacaine injection
- Sham SGB (Placebo Comparator): One time administration
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ropivacaine injection — 6.5cc of Ropivacaine hydrochloride (HCl) 0.5%, one time into the stellate ganglion
  Other Names: Naropin
  Arms: Stellate Ganglion Block
Drug: Normal saline — 6.5cc of Normal Saline one time into the stellate ganglion.
  Arms: Sham SGB

SUMMARY:
The goal of this clinical trial is to compare the combination of Massed Prolonged Exposure (PE); a behavioral therapy for PTSD) and a stellate ganglion block (SGB; an injection of a local anesthetic into the front of the neck) with Massed Prolonged Exposure and a sham injection in a sample of military service members or retirees with PTSD. The main questions it aims to answer are: (1) Does the addition of an SGB improve treatment outcomes associated with Massed PE and (2) Do differences in psychophysiological arousal during the exposure portion of treatment help explain treatment outcomes for PTSD. Participants will receive ten 90-minute session of Massed PE. Between the first and second Massed PE sessions, half of the participants will receive a SGB, and half will receive a sham SGB.

DETAILED DESCRIPTION:
Massed PE will be conducted by master-level or doctoral-level therapists. Participants will meet with their providers for individual, 90-minute sessions. They will then be asked to complete out-of-session treatment assignments throughout the rest of the day. Between the individual therapy session and out-of-session treatment assignments, participants will engage in approximately four to six hours of treatment per day, Monday through Friday, for two weeks. Each participant will also be offered three booster sessions at 1-, 3-, and 7-weeks posttreatment.

The stellate ganglion block injection or the sham SGB will be administered between the first and second massed PE session by qualified medical personnel as per standard operating procedure for the placement of a stellate ganglion block. A research nurse will be in attendance during the procedure and for an hour recovery period following the block administration.

Assessments will be administered at pretreatment, during treatment, at posttreatment, and at 1-, 3-, and 6-months following the completion of PE. The primary outcome assessment will be 1-month following the completion of PE. Following this assessment, participants randomized to the sham SGB arm of the study will be offered an SGB with ropivacaine.

ELIGIBILITY:
Inclusion Criteria:

1. Active duty and retired military service members ages 18-65 years
2. PTSD diagnosis as assessed by Clinician-Administered Posttraumatic Stress Scale
3. Able to speak and read English (due to standardization of outcome measures)
4. Defense Enrollment Eligibility Reporting System (DEERS)-eligible to receive care at a military treatment facility (MTF) where the stellate ganglion block will be placed.

Exclusion Criteria:

1. Current suicidal ideation severe enough to warrant immediate attention (as determined by the Depressive Symptoms Index - Suicidality Subscale and the Self-Injurious Thoughts and Behaviors Interview short form) and corroborated by a clinical risk assessment by a credentialed provider.
2. Current manic episode or psychotic symptoms requiring immediate stabilization or hospitalization (as determined by clinical judgment)
3. Symptoms of moderate to severe substance use (to include alcohol) warranting immediate intervention based on clinical judgment.
4. Other psychiatric disorders severe enough to warrant designation as the primary disorder as determined by clinician judgment
5. Pregnancy or breastfeeding
6. Current anticoagulant use
7. History of bleeding disorder
8. Infection or mass at injection site
9. Myocardial infarction within 6 months of procedure
10. Pathologic bradycardia or irregularities of heart rate or rhythm
11. Symptomatic hypotension
12. Phrenic or laryngeal nerve palsy
13. History of glaucoma
14. Uncontrolled seizure disorder
15. History of allergy to local anesthetics
16. Current use of Class III antiarrhythmics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Clinician-Administered PTSD Scale-DSM 5 (CAPS-5) | Baseline and at 1-month, 3-month, and 6-month follow-up assessments
  A 30-item structured interview used to assess change symptoms of PTSD. Questions target the onset and duration of symptoms, subjective distress, impact on social and occupational functioning. Total severity scores range from 0 to 80 with higher score indicative of greater PTSD severity. The measure can also be used to confirm the presence of a PTSD diagnosis.
Change from baseline in Posttraumatic Stress Disorder Checklist -DSM 5 (PCL-5) | Baseline and at 1-month, 3-month, and 6-month follow-up assessments
  A 20-item self-report measure that assesses the presence and change in severity of PTSD symptoms using the Diagnostic and Statistical Manual of mental disorders (DSM-5). Total severity scores range from 0 to 80 with higher score indictive of greater PTSD severity.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 items (PHQ-9) | Baseline and at 1-month, 3-month, and 6-month follow-up assessments
  A 9-item self-report measure that assesses the presence and change in severity of depressive symptoms. Total scores range from 0 to 27 with higher scores reflective of greater severity.
General Anxiety Disorder Screener - 7 Items (GAD-7) | Baseline and at 1-month, 3-month, and 6-month follow-up assessments
  A 9-item self-report measure that assesses the presence and change in severity of general anxiety symptoms. Total scores range from 0 to 21 with higher scores reflective of greater severity.
Posttraumatic Cognitions Inventory (PTCI) | Baseline and at 1-month, 3-month, and 6-month follow-up assessments
  A 36-item self-report measure that assesses change in self-blame, negative cognitions about self, and negative cognitions about the world following trauma exposure. Total scores range from 33 to 231 with higher scores reflective of more problematic cognitions.
Psychophysiological arousal - Galvanic Skin Response | Two weeks
  Change in Psychophysiological data collected from a smart watch measuring galvanic skin response
Psychophysiological arousal - Skin Temperature | Two weeks
  Change in Psychophysiological data collected from a smart watch measuring skin temperature
Psychophysiological arousal - Heart Rate | Two weeks
  Change in Psychophysiological data collected from a smart watch measuring heart rate
Psychophysiological arousal - Interbeat Interval | Two weeks
  Change in Psychophysiological data collected from a smart watch measuring interbeat interval
Psychophysiological arousal - Three-Dimensional Accelerometer Movement | Two weeks
  Change in Psychophysiological data collected from a smart watch measuring three-dimensional accelerometer movement
Psychophysiological arousal - Electrodermal Activity | Two weeks
  Change in Psychophysiological data collected from a smart watch measuring electrodermal activity
Psychophysiological arousal - Photoplethysmography | Two weeks
  Change in Psychophysiological data collected from a smart watch measuring photoplethysmography

CONTACTS AND LOCATIONS:
Overall Officials: Alan Peterson, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - Carl R. Darnall Army Medical Center, Fort Hood, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foa EB, McLean CP, Zang Y, Rosenfield D, Yadin E, Yarvis JS, Mintz J, Young-McCaughan S, Borah EV, Dondanville KA, Fina BA, Hall-Clark BN, Lichner T, Litz BT, Roache J, Wright EC, Peterson AL; STRONG STAR Consortium. Effect of Prolonged Exposure Therapy Delivered Over 2 Weeks vs 8 Weeks vs Present-Centered Therapy on PTSD Symptom Severity in Military Personnel: A Randomized Clinical Trial. JAMA. 2018 Jan 23;319(4):354-364. doi: 10.1001/jama.2017.21242. PMID 29362795
- [Background] Hanling SR, Hickey A, Lesnik I, Hackworth RJ, Stedje-Larsen E, Drastal CA, McLay RN. Stellate Ganglion Block for the Treatment of Posttraumatic Stress Disorder: A Randomized, Double-Blind, Controlled Trial. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):494-500. doi: 10.1097/AAP.0000000000000402. PMID 27187898
- [Background] Lipov EG, Joshi JR, Lipov S, Sanders SE, Siroko MK. Cervical sympathetic blockade in a patient with post-traumatic stress disorder: a case report. Ann Clin Psychiatry. 2008 Oct-Dec;20(4):227-8. doi: 10.1080/10401230802435518. No abstract available. PMID 19034755
- [Background] Lynch JH, Mulvaney SW, Kim EH, de Leeuw JB, Schroeder MJ, Kane SF. Effect of Stellate Ganglion Block on Specific Symptom Clusters for Treatment of Post-Traumatic Stress Disorder. Mil Med. 2016 Sep;181(9):1135-41. doi: 10.7205/MILMED-D-15-00518. PMID 27612365
- [Background] Mulvaney SW, Lynch JH, Hickey MJ, Rahman-Rawlins T, Schroeder M, Kane S, Lipov E. Stellate ganglion block used to treat symptoms associated with combat-related post-traumatic stress disorder: a case series of 166 patients. Mil Med. 2014 Oct;179(10):1133-40. doi: 10.7205/MILMED-D-14-00151. PMID 25269132
- [Background] Odosso RJ, Petta L. The Efficacy of the Stellate Ganglion Block as a Treatment Modality for Posttraumatic Stress Disorder Among Active Duty Combat Veterans: A Pilot Program Evaluation. Mil Med. 2021 Jul 1;186(7-8):e796-e803. doi: 10.1093/milmed/usaa246. PMID 33242072
- [Background] Peterson AL, Blount TH, Foa EB, Brown LA, McLean CP, Mintz J, Schobitz RP, DeBeer BR, Mignogna J, Fina BA, Evans WR, Synett S, Hall-Clark BN, Rentz TO, Schrader C, Yarvis JS, Dondanville KA, Hansen H, Jacoby VM, Lara-Ruiz J, Straud CL, Hale WJ, Shah D, Koch LM, Gerwell KM, Young-McCaughan S, Litz BT, Meyer EC, Blankenship AE, Williamson DE, Roache JD, Javors MA, Sharrieff AM, Niles BL, Keane TM; Consortium to Alleviate PTSD. Massed vs Intensive Outpatient Prolonged Exposure for Combat-Related Posttraumatic Stress Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jan 3;6(1):e2249422. doi: 10.1001/jamanetworkopen.2022.49422. PMID 36602803